CLINICAL TRIAL: NCT04379375
Title: Using Behavioral Nudges to Improve Preventive Health Behaviors That Limit COVID-19 Spread
Brief Title: Nudges to Improve Health Behaviors That Limit COVID-19 Spread
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment rate
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Advancing a Healthier Wisconsin Endowment (Unknown)
Responsible Party: Principal Investigator, Nicholas D. Young, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00037864
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Health Behavior; COVID-19
MeSH Terms: conditions — Health Behavior; COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inertia (Active Comparator): Participants simply receive and subsequently have "default" access (i.e., readily and immediately available) to handwashing (HW) materials. This condition will functionally serve as a control comparison. As the term implies, inertia capitalizes on minimizing effort necessary (e.g., going to the grocery store) to engage in HW behavior in one's personal environment.
  Interventions: Behavioral: Nudge
- Anchoring (Experimental): Involves once again providing "default access" to HW materials as above, but adds an explicit written cue to wash hands at a rate of (15) times per day, which is placed directly on the soap dispenser. The stimulus is intended to deliberately prime participant thinking (and subsequent behavior) towards a higher reference point that "overshoots" a desired target rate of 10+ daily HWs.
  Interventions: Behavioral: Nudge

INTERVENTIONS:
Behavioral: Nudge — Application of behavior-change strategies based on principles of behavioral economics, decision-making heuristics, psychological/environmental variables.

SUMMARY:
This investigation is a randomized intervention trial that evaluates behavioral nudges (BN) to increase hand washing behavior and subsequently reduce COVID-19 spreading to a targeted high-risk patient population based in Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Provision of signed and dated informed consent form
* Willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Has at least 1 risk factor associated with COVID-19 documented in their electronic medical record
* Followed by (i.e., actively receiving care) from targeted MCW specialties (Internal Medicine, OBGYN, Surgery)
* Access to necessary resources for participating in a technology-based activities (i.e., internet access + mobile phone or computer to complete online survey)
* Maintains a personal address where study materials can be shipped and where participant lives full time

Exclusion Criteria:

* Previous COVID-19 diagnosis or positive COVID-19 test result documented in their electronic medical record
* Current participation in another treatment or intervention study associated with COVID-19
* Previous documented Obsessive-Compulsive Disorder diagnosis in their electronic medical record
* Non-English speaker
* Patients hospitalized or incapacitated at onset of potential enrollment
* No access to electronic platform with internet (e.g., smartphone, tablet, computer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Hand Washing Behavior | 8 weeks post-enrollment
  Measured via adapted version of a previously validated questionnaire (Hygiene Inventory - 23), which specifically includes (a) 1 item about approximate hand washing frequency on an average day, with response options of whole numbers from 0-29 and an additional option of "30 or more" where higher numbers are generally considered better outcomes, (b) 10 items about hand washing behavior in various contexts, with response options of "1 - Never", "2 - Occasionally", "3 - Usually", and "4 - Always" where higher scores are considered better outcomes, and (c) 1 item about general hand hygiene using antibacterial gel or wipes, with response options of "1 - Never", "2 - Occasionally", "3 - Usually", and "4 - Always" where higher scores are considered better outcomes.

SECONDARY OUTCOMES:
Clinical Outcomes - General/Internal Medicine | 12 weeks post-enrollment
  Patient frequency/rate for the following variables measured via electronic medical record:
  ED visit (respiratory illness/other) ED visit reason (if non-respiratory) Admission (respiratory Illness) Respiratory Illness secondary to COVID19 ICU admission due to respiratory illness ICU admission due to COVID19 Mechanical Respiratory support Duration of Mechanical support (days) Mortality (respiratory Illness/other)
Clinical Outcomes - Obstetrics & Gynecology | 12 weeks post-enrollment
  Patient frequency/rate for the following variables measured via electronic medical record:
  Respiratory Illness at time of Delivery Pre-delivery COVID19 testing Delivery plan altered due to respiratory illness Miscarriage Preterm labor/birth Preeclampsia Respiratory Illness in newborn Newborn COVID19 testing
Clinical Outcomes - Surgery | 12 weeks post-enrollment
  Patient frequency/rate for the following variables measured via electronic medical record:
  Respiratory Illness at time of surgery Pre-Operative COVID19 testing Surgery delayed due to respiratory illness Surgery delayed due to COVID19 positive Adverse outcome secondary to delay in surgery Post operative intubation >2 days Post operative unplanned reintubation Post operative pneumonia Post operative respiratory illness secondary to COVID19

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D Young, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No